CLINICAL TRIAL: NCT01560429
Title: Efficacy of Patient Controlled Epidural Anesthesia (PCEA) Versus Continuous Epidural Analgesia (CEA) for Post-thoracotomy Pain.
Brief Title: Efficacy of Patient Controlled Epidural Anesthesia Versus Continuous Epidural Analgesia for Post-thoracotomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Vidur Shyam, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANAE-147-08; ANAE-147-08 (Other: Queens University REB)
Record Dates: First submitted 2012-03-06; First posted 2012-03-22 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Acute Post-thoracotomy Pain
Keywords: anesthesia and analgesia; Epidural Anesthesia; administration schedules, drug
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient controlled epidural analgesia (Experimental): An epidural catheter sited preoperatively so analgesics can be administered postoperatively. Patients were titrated on a continuous analgesic epidural infusion until stable pain scores of ≤ 3 were reached while in PACU. Once stable, they were allocated to their preoperatively determined randomization which meant they still received 2/3rd of the anesthetic as a background infusion but also had the option to self-administer the remaining 1/3rd dose as patient controlled epidural analgesia (PCEA). Rescue analgesia was available upon request.
  Interventions: Procedure: Patient controlled epidural analgesia
- continuous epidural analgesia (Active Comparator): An epidural catheter sited preoperatively so analgesics can be administered postoperatively. Patients were titrated on a continuous analgesic epidural infusion rate until stable pain scores of ≤ 3 were reached while in PACU (as described in the PCEA group). Once stable, they were allocated to their preoperatively determined randomization assignment which for the CEA group meant they remained on the continuous background epidural infusion rate previously determined to maintain pain scores ≤ 3 while in PACU. Rescue analgesia was available as needed.
  Interventions: Procedure: Continuous epidural analgesia

INTERVENTIONS:
Procedure: Patient controlled epidural analgesia — Continuous epidural infusion rates were set to maintain pain scores of ≤ 3 on a numeric rating scale (NRS) of 0 to 10 while in the post anesthesia care unit (PACU) following thoracotomy. Once stabilized patients were switched to Patient controlled epidural analgesia (PCEA) which meant they continued to receive 2/3rds of the dose as continuous background epidural infusions but they had the option to receive the remaining 1/3rd dosage via PCEA.
  Other Names: PCEA
  Arms: Patient controlled epidural analgesia
Procedure: Continuous epidural analgesia — The continuous epidural analgesia (CEA) infusion rates were titrated to achieve pain scores of ≤ 3 on a numeric rating scale (NRS) of 0 to 10 while in post-anesthesia care unit (PACU) (as described for the PCEA group above). Those allocated to the CEA group remained on the same continuous epidural analgesia infusion which maintained the pain scores at ≤ 3.
  Other Names: CEA
  Arms: continuous epidural analgesia

SUMMARY:
Postoperative thoracotomy pain is normally managed with an epidural catheter and continuous epidural analgesia (CEA). However, for some surgical procedures, patient controlled epidural anesthesia (PCEA) is more effective but little research has compared the two methods following thoracotomy. The current randomized, prospective clinical investigation did just this. Following institutional ethics approval 52 patients scheduled for thoracotomy were recruited for this prospective, randomized, unblinded study. A thoracic epidural catheter was sited preoperatively. Postoperatively all patients were titrated on continuous epidural infusions (hydromorphone 10 mcg/mL + bupivacaine 1 mg/mL) until pain scores were stable at ≤3 on a numeric rating scale (NRS). Then they were allocated to their preoperatively determined randomization (either remained on continuous epidural infusion or they were switched to receive 2/3 of the stabilized background dose via continuous epidural infusion with the option to self-administer the remaining 1/3rd of the dose via PCEA. Participants remained on their allocated analgesic regimens for 48 hours postoperatively. The primary outcome was consumption of local anaesthetics/opioids. The secondary outcomes were worst pain and pain while coughing (0-10 NRS).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* American Society of Anesthesiologist's (ASA) Physical Status I-III
* Body Mass Index (BMI) < 40
* Able to use a PCEA device

Exclusion Criteria:

* Intolerance/hypersensitivity to agents used in the study
* Contraindication to epidural placement
* Current alcohol/substance abuse
* Chronic pain condition requiring chronic analgesic
* BMI ≥ 40 or body weight less than 50kg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vidur Shyam, MBBS, FRCPC, Principal Investigator — Queen's University & Kingston General Hospital
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled prior to thoracotomy. 52 patients were randomized to receive PCEA (n=26) or CEA (n=26).
Groups:
- Patient-controlled Epidural Analgesia: All patients were preoperatively sited with an epidural catheter in preparation for postoperative pain management. Continuous epidural infusion rates were set to achieve scores of ≤ 3 on a numeric rating scale (NRS) of 0 to 10 while in PACU. Upon allocation to the preoperatively determined randomization, the PCEA were switched the receive 2/3 of their baseline infusion as continuous background infusion but they also had the option to self administered the remaining 1/3rd of the dose via patient controlled epidural analgesia (PCEA)
- Continuous Epidural Analgesia: All patients were preoperatively sited with an epidural catheter in preparation for postoperative pain management. Postoperatively all patients received continuous epidural analgesia at infusion rates to reach pain scores of ≤ 3 while in PACU. Those randomized to the Continuous epidural analgesia group remained on the same CEA regimen.
Period: Overall Study
Arm/Group | Patient-controlled Epidural Analgesia | Continuous Epidural Analgesia
Started | 26 | 26
Completed | 23 | 20
Not Completed | 3 | 6
Not completed — Protocol Violation | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Patient-controlled Epidural Analgesia: All patients were preoperatively sited with an epidural catheter in preparation for postoperative pain management. Patient controlled epidural analgesia : CEA infusion rates were set when pain scores of ≤ 3 on a numeric rating scale (NRS) of 0 to 10 were achieved in the post-anesthesia care unit (PACU). Continuous epidural analgesia : PCEA parameters were adjusted to allow an equivalent dose per hour.
- Continuous Epidural Analgesia: All patients were preoperatively sited with an epidural catheter in preparation for postoperative pain management. Patient controlled epidural analgesia : CEA infusion rates were set when pain scores of ≤ 3 on a numeric rating scale (NRS) of 0 to 10 were achieved in PACU. Continuous epidural analgesia : PCEA parameters were adjusted to allow an equivalent dose per hour.
- Total: Total of all reporting groups
Arm/Group | Patient-controlled Epidural Analgesia | Continuous Epidural Analgesia | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years]
  Between 18 and 65 years | 60.8 (5.2) | 56.7 (5.9) | 58 (5.9)
  >=65 years | 70.9 (4.1) | 70.6 (3.1) | 70.8 (3.6)
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (6.1) | 62.7 (8.5) | 65.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Local Anesthetic Consumption
Description: Amount of anesthetic consumed (either through epidural catheter or as rescue bolus at 48 hours following thoracotomy administered either through CEA or PCEA.
Time Frame: 48 hours postoperatively
Measure: Mean (Standard Error); unit: ug
Groups:
- Patient-controlled Epidural Analgesia: An epidural catheter sited preoperatively so analgesics can be administered postoperatively. Patients were titrated on a continuous analgesic epidural infusion until stable pain scores of ≤ 3 were reached while in PACU. Once stable, they were allocated to their preoperatively determined randomization which meant they still received 2/3rd of the anesthetic as a background infusion but also had the option to self-administer the remaining 1/3rd dose as patient controlled epidural analgesia (PCEA). Rescue analgesia was available upon request.
- Continuous Epidural Analgesia: All patients were preoperatively sited with an epidural catheter in preparation for postoperative pain management. CEA infusion rates were set to achieve pain scores of ≤ 3 on a numeric rating scale (NRS) of 0 to 10 while in PACU. Those allocated to the CEA group remained on the same continuous epidural infusion rate to which they were optimized.
Arm/Group | Patient-controlled Epidural Analgesia | Continuous Epidural Analgesia
Number analyzed (Participants) | 23 | 20
ug | 1505.39 (339.43) | 1862.16 (493.85)

2. Secondary Outcome: Worst Pain Scores
Description: worst pain scores on numerical rating scale (0-10, where 10 is the worst) at 24 & 48 hours following surgery
Time Frame: 48 hours postoperatively
Reporting Status: Not Posted

3. Secondary Outcome: Worst Pain While Coughing
Description: Worst pain on a numerical rating scale(0-10 worst) at 24 and 48 hours following thoracotomy
Time Frame: 48 hours postoperatively
Reporting Status: Not Posted

4. Primary Outcome: Anesthetic Consumption (mg)
Description: amount of anesthetic consumed was calculated for each group over time.
Time Frame: 4,8,12, 24 and 48 hours postoperatively
Measure: Mean (Standard Error); unit: mg
Groups:
- Patient-controlled Epidural Analgesia; Continuous Epidural Analgesia: All patients were preoperatively sited with an epidural catheter in preparation for postoperative pain management. Patient controlled epidural analgesia : CEA infusion rates were set when pain scores of ≤ 3 on a numeric rating scale (NRS) of 0 to 10 were achieved in PACU. Continuous epidural analgesia : PCEA parameters were adjusted to allow an equivalent dose per hour.
Arm/Group | Patient-controlled Epidural Analgesia | Continuous Epidural Analgesia
Number analyzed (Participants) | 23 | 20
mg | 158.9 (73.5) | 181.5 (73.5)

ADVERSE EVENTS:
Arm/Group | Patient-controlled Epidural Analgesia | Continuous Epidural Analgesia
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes